CLINICAL TRIAL: NCT05070702
Title: First in Human Study in Healthy Subjects to Investigate the Safety, Tolerability and Pharmacokinetics of Single Ascending and Repeat Doses of CT-1500
Brief Title: First in Human Study of CT-1500 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Circadian Therapeutics Ltd (Industry)
Collaborators: Neuroscience Trials Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: CT-1500-01
Record Dates: First submitted 2021-09-13; First posted 2021-10-07 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Ascending Single Doses followed by Ascending Multiple Doses of Study Intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active and Placebo capsules are identical in appearance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CT-1500 Active (SAD) (Experimental): 6 out of 8 participants per cohort (up to 5 cohorts) will be randomized to receive a single oral dose of CT-1500 between 5 mg and 120 mg
  Interventions: Drug: CT-1500
- Placebo (SAD) (Placebo Comparator): 2 out of 8 participants per cohort (up to 5 cohorts) will be randomized to receive a single oral dose of matching placebo
  Interventions: Drug: Placebo
- CT-1500 Active (MAD) (Experimental): 6 out of 8 participants per cohort (up to 3 cohorts) will be randomized to receive 7 daily oral doses of CT-1500 between 5 and 45 mg
  Interventions: Drug: CT-1500
- Placebo (MAD) (Placebo Comparator): 2 out of 8 participants per cohort (up to 3 cohorts) will be randomized to receive 7 daily oral doses of matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT-1500 — Hard Capsule
  Arms: CT-1500 Active (MAD); CT-1500 Active (SAD)
Drug: Placebo — Hard Capsule
  Arms: Placebo (MAD); Placebo (SAD)

SUMMARY:
This study is a single center, randomized, placebo-controlled, double-blind study of CT-1500 in healthy volunteers. The study will evaluate the safety, tolerability and pharmacokinetics of single ascending doses and multiple ascending doses of orally administered CT-1500 compared to placebo.

DETAILED DESCRIPTION:
This study is a single center, randomized, placebo-controlled, double-blind study of CT-1500 in healthy volunteers. The study will evaluate the safety, tolerability and pharmacokinetics of single ascending doses and multiple ascending doses of orally administered CT-1500 compared to placebo. It is planned for 5 dose levels to be investigated in the single ascending dose (SAD) part (Part 1) of the study, between 5 mg to 120 mg. Three dose levels are proposed for investigation in the multiple ascending dose (MAD) part (Part 2) of the study.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy with the exception of those medical conditions allowed per the study criteria
* Able to provide voluntary, written informed consent with comprehension of all aspects of the protocol, prior to any study procedures
* Body Mass Index (BMI) of 18.5 to 32 kg/m2 and weight >48 kg
* Systolic Blood Pressure (BP) of 90-140 mmHg, Diastolic BP of 40-90 mmHg and Heart Rate between 40 and 100 bpm
* Forced Expiratory Volume in one second (FEV1) > 85% predicted
* Clinical laboratory results at screening and Day -1 to be within normal limits unless deemed as not clinically significant by the investigator
* Willing to consume bovine containing products (investigational product capsules are bovine gelatin in origin);
* Agree not to donate blood or plasma products for at least 30 days after the end of study (EOS) visit
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at Day -1, must not be breastfeeding, lactating or planning a pregnancy and must use an acceptable form of contraception during the treatment period and for 32 days after the last dose
* Male participants with a female partner of childbearing potential must agree to use an acceptable form of contraception during the treatment period and for 92 days after the last dose

Exclusion Criteria:

* Significant current or historical disease, including intercurrent illness in the 4 weeks prior to screening
* Current or historical diagnosis of sleep disorders
* Hepatic disorders other than benign unconjugated hyperbilirubinaemia
* History of moderate or severe psychiatric illness
* History of severe allergy or anaphylaxis to any drug, food, toxin or other exposure
* Heavy caffeine drinker in the last 3 months. If subjects are willing to reduce their caffeine intake for 14 days prior to first dose and for the duration of the study, they can participate
* Hypersensitivity to CT-1500 or any of the inert excipients in the capsule formulation
* Positive hepatitis B surface antigen (HBsAg), positive hepatitis C antibody (HCV) or positive human immunodeficiency virus (HIV) test
* Treatment with an investigational drug within 30 days or less than 5 half-lives (whichever is longer) prior to screening
* Use of prescription medication within 14 days prior to investigational product administration until the end of study visit, with the exception of oral contraceptives.
* Use of over-the-counter medication and supplements for 7 days prior to investigation product administration until the end of study visit. Exceptions at the discretion of the investigator.
* Receipt of a Coronavirus disease 2019 (COVID-19) vaccine within 14 days prior to investigational product administration or a planned second dose of a COVID-19 vaccine during study participation
* Use of tobacco or nicotine-containing products in excess of 2 cigarettes per day within 1 month prior to screening
* Major surgery in the 6 months preceeding screening or planned surgery during the study
* Donated blood or blood products or had a substantial loss of blood with 3 months prior to screening
* A history of drug abuse or addiction
* A history of alcoholism or consumption of more than 3 alcoholic drinks per day or consumption of alcohol within 48 hours prior to first dose
* Unable to abstain from grapefruit-containing foods or beverages or Seville orange-containing foods or beverages from 48 hours prior to investigational product administration until completion of the confinement period;
* Unable to avoid heavy exercise (eg, marathon runners, weight-lifters) from 48 hours prior to investigational product administration until completion of the confinement period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) during the SAD part of the study | Initiation of dosing through 7 days post dose
  Incidence and severity of AEs and SAEs
Adverse Events and Serious Adverse Events during the MAD part of the study | Initiation of dosing through 14 days post dose
  Incidence and severity of AEs and SAEs
Tolerability of CT-1500 as defined by change from baseline in Heart Rate (SAD) | Initiation of dosing through 7 days post dose
Tolerability of CT-1500 as defined by change from baseline in Heart Rate (MAD) | Initiation of dosing through 14 days post dose
Tolerability of CT-1500 as defined by change from baseline in Respiratory Rate (SAD) | Initiation of dosing through 7 days post dose
Tolerability of CT-1500 as defined by change from baseline in Respiratory Rate (MAD) | Initiation of dosing through 14 days post dose
Tolerability of CT-1500 as defined by change from baseline in Electrocardiogram Assessment (SAD) | Initiation of dosing through 7 days post dose
  Change in QT interval from baseline
Tolerability of CT-1500 as defined by change from baseline in Electrocardiogram assessment (MAD) | Initiation of dosing through 14 days post dose
  Change in QT interval from baseline
Tolerability of CT-1500 as defined by change from baseline in Spirometry assessment (SAD) | Initiation of dosing through 7 days post dose
  Change from baseline in Forced Expiratory Volume in 1 second (FEV1)
Tolerability of CT-1500 as defined by change from baseline in Spirometry assessment (MAD) | Initiation of dosing through 14 days post dose
  Change from baseline in Forced Expiratory Volume in 1 second (FEV1)
Change in Renal function from baseline (SAD) | Initiation of dosing through 24 hours post dose
  Renal Function as assessed by change in estimated Glomerular Filtration Rate from baseline
Change in Renal function from baseline (MAD) | Initiation of dosing on Day 1 through 24 hours and initiation of dosing on Day 7 through 24 hours
  Renal Function as assessed by change in estimated Glomerular Filtration Rate from baseline

SECONDARY OUTCOMES:
Pharmacokinetic parameter: AUC-last (SAD) | Baseline (predose) through 48 hours post dose
  Area under the plasma concentration time curve (AUC) from time zero until the last measurable concentration of CT-1500 is observed during the SAD part of the study
Pharmacokinetic parameter: AUC-last (SAD) | Baseline (predose) through 48 hours post dose
  Area under the plasma concentration time curve from time zero until the last measurable concentration of metabolite CT-1517 is observed during the SAD part of the study
Pharmacokinetic parameter: AUC-last (SAD) | Baseline (predose) through 48 hours post dose
  Area under the plasma concentration time curve from time zero until the last measurable concentration of metabolite CT-1518 is observed during the SAD part of the study
Pharmacokinetic parameter: AUC-last (MAD) | Baseline (predose) on Day 1 through 24 hours post dose and Baseline (predose) on Day 7 through 24 hours
  Area under the plasma concentration time curve from time zero until the last measurable concentration of CT-1500 is observed during the MAD part of the study
Pharmacokinetic parameter: AUC-last (MAD) | Baseline (predose) on Day 1 through 24 hours post dose and Baseline (predose) on Day 7 through 24 hours
  Area under the plasma concentration time curve from time zero until the last measurable concentration of metabolite CT-1517 is observed during the MAD part of the study
Pharmacokinetic parameter: AUC-last (MAD) | Baseline (predose) on Day 1 through 24 hours post dose and Baseline (predose) on Day 7 through 24 hours
  Area under the plasma concentration time curve from time zero until the last measurable concentration of metabolite CT-1518 is observed during the MAD part of the study
Pharmacokinetic parameter: AUC-inf (SAD) | Baseline (predose) through 48 hours post dose
  Area under the plasma concentration time curve from time zero to infinity of CT-1500 is observed during the SAD part of the study
Pharmacokinetic parameter: AUC-inf (MAD) | Baseline (predose) on Day 1 through 24 hours post dose and Baseline (predose) on Day 7 through 24 hours
  Area under the plasma concentration time curve from time zero to infinity of CT-1500 is observed during the MAD part of the study
Pharmacokinetic parameter: Cmax (SAD) | Baseline (predose) through 48 hours post dose
  Maximal measured plasma concentration (Cmax) of CT-1500 during the SAD part of the study
Pharmacokinetic parameter: Cmax (SAD) | Baseline (predose) through 48 hours post dose
  Maximal measured plasma concentration of metabolite CT-1517 during the SAD part of the study
Pharmacokinetic parameter: Cmax (SAD) | Baseline (predose) through 48 hours post dose
  Maximal measured plasma concentration of metabolite CT-1518 during the SAD part of the study
Pharmacokinetic parameter: Cmax (MAD) | Baseline (predose) on Day 1 through 24 hours post dose and Baseline (predose) on Day 7 through 24 hours
  Maximal measured plasma concentration of CT-1500 during the MAD part of the study
Pharmacokinetic parameter: Cmax (MAD) | Baseline (predose) on Day 1 through 24 hours post dose and Baseline (predose) on Day 7 through 24 hours
  Maximal measured plasma concentration of metabolite CT-1517 during the MAD part of the study
Pharmacokinetic parameter: Cmax (MAD) | Baseline (predose) on Day 1 through 24 hours post dose and Baseline (predose) on Day 7 through 24 hours
  Maximal measured plasma concentration of metabolite CT-1518 during the MAD part of the study
Pharmacokinetic parameter: Tmax (SAD) | Baseline (predose) through 48 hours post dose
  Time when Maximal measured plasma concentration is observed (Tmax) of CT-1500 during the SAD part of the study
Pharmacokinetic parameter: Tmax (SAD) | Baseline (predose) through 48 hours post dose
  Time when Maximal measured plasma concentration is observed of metabolite CT-1517 during the SAD part of the study
Pharmacokinetic parameter: Tmax (SAD) | Baseline (predose) through 48 hours post dose
  Time when Maximal measured plasma concentration is observed of metabolite CT-1518 during the SAD part of the study
Pharmacokinetic parameter: Tmax (MAD) | Baseline (predose) on Day 1 through 24 hours post dose and Baseline (predose) on Day 7 through 24 hours
  Time when Maximal measured plasma concentration is observed of CT-1500 during the MAD part of the study
Pharmacokinetic parameter: Tmax (MAD) | Baseline (predose) on Day 1 through 24 hours post dose and Baseline (predose) on Day 7 through 24 hours
  Time when Maximal measured plasma concentration is observed of metabolite CT-1517 during the MAD part of the study
Pharmacokinetic parameter: Tmax (MAD) | Baseline (predose) on Day 1 through 24 hours post dose and Baseline (predose) on Day 7 through 24 hours
  Time when Maximal measured plasma concentration is observed of metabolite CT-1518 during the MAD part of the study

CONTACTS AND LOCATIONS:
Overall Officials: Philip Ryan, Dr, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The Sponsor will consider requests from appropriately qualified researchers for study information and participant data upon a formal request to contact@circadiantherapeutics.com.
Supporting Information: Study Protocol, CSR